CLINICAL TRIAL: NCT01142453
Title: Therapy Optimisation Using High-frequency and High-dosage Administration of Interferon-beta (Rebif®) in MS Patients. Case Series for Adjustment of Treatment Strategy and Its Monitoring
Brief Title: An Observational Study Evaluating Therapy Optimisation Using High-frequency and High-dosage Administration of Interferon-beta (Rebif®) in Multiple Sclerosis (MS) Patients
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Gesellschaft für Therapieforschung mbH (Industry)
Responsible Party: Dr. Norbert Zessack/Head of Medicine BU Neurology, Merck Serono GmbH Germany, an affiliate of MerckKGaA, Darmstadt, Germany
Other Study IDs: HDHF PMS
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2010-06

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Multiple sclerosis; Rebif; Interferon
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood

INTERVENTIONS:
Drug: Interferon beta 1a — A dosage of 44 µg interferon beta 1a subcutaneous self-injection three times a week was recommended for therapy of the included, suitable MS subjects after a creep-in phase (depending on the respective preliminary therapy)
  Other Names: Rebif

SUMMARY:
This was an observational, single arm, multicentric study conducted for the adjustment of treatment strategy and its monitoring using high-frequency and high-dosage administration of interferon-beta (Rebif) in MS subjects. Study focussed on assessment of the effectiveness and safety of existing immunomodulatory basis therapy in MS subjects.

DETAILED DESCRIPTION:
Treatment of MS, which progresses to attacks or episodes, with interferon-beta has established itself as therapy of the first choice. On the basis of different studies, the hypothesis was substantiated that the effectiveness is dependent on dose and application frequency. These realizations justify the use of high-dose interferon-beta not only in subjects in the initial stages of disease, but also in those subjects, who have a progressing disease activity even in the advanced stage, if other therapies fail. For achieving maximum benefit for the subject, an optimum therapy is imperative. The therapy plan (Immunomodulatory Therapy) of "MS Therapy Consensus Group" (MSTKG) is being widely used. In the article: "Optimising lmmunomodulatory Therapy for MS Patients" that appeared in the "International Journal of MS care" in the year 2002, a simple 9-scale model" is proposed that defines four areas respectively: not conspicuous, conspicuous, alarming and measures are necessary, in the three areas: attacks/episodes, disease progression and magnetic resonance tomography (MRT). The modification of an existing therapy, such as modifying the application plan, increasing the dosage, or substance change is recommended, if 'conspicuousness' is shown in all three areas, two areas are shown as 'alarming' or an area is shown as 'action necessary'. The decision for a therapy adjustment with the help of the "three scale model" should not happen solely on the results of the MRT. The model in the study involved attack or episode pertaining to: frequency, degree of severity, ability of involution and the response to a cortisone pulse therapy.

OBJECTIVES

* To assess the effectiveness and safety of existing immunomodulatory basis therapy in MS subjects
* To identify candidates suitable for possible therapy adjustment

ELIGIBILITY:
Inclusion Criteria:

* Subjects with clinically ensured diagnosis of a MS and history of attacks or episodes
* Subjects who were on one of the permitted basis therapies at least since 6 months
* Subjects with existing systemic concurrent diseases (e.g.diabetes, heart, liver, kidney diseases) should be monitored very carefully.

Exclusion Criteria:

* Subjects with secondary progressive course of the MS without attacks or episodes, pregnant or nursing subjects as well as subjects with history of contraindications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with clinically ensured diagnosis and history of attacks or episodes of a MS and on one of the permitted basis therapies at least since 6 months were enrolled for the case series
Sampling Method: Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2005-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The course of the therapy, the assessment of the effectiveness, safety and compatibility were documented over the observation period | Beginning to 12 months observation period
  Subject's therapy status was assessed with the help of a ready-made evaluation sheet, modified according to the so-called "Scale Model"

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Norbert Zessack, Study Director — Merck Serono GmbH, Germany